CLINICAL TRIAL: NCT01687920
Title: Single Center, Randomized, Open-label, 5-fold Crossover Study in Healthy Male Subjects to Investigate the Pharmacokinetic Dose Proportionality of BAY94-8862 Given as 5 Different Single Oral IR Tablet Doses (1.25, 2.5, 5.0, 7.5 and 10 mg)
Brief Title: Dose Proportionality Study With BAY94-8862 IR (Immediate Release) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15481; 2012-003055-10 (EudraCT Number)
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
Keywords: Cardiac disorders
MeSH Terms: conditions — Heart Failure; Heart Diseases | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- BAY94-8862 (1.25mg) (Experimental): single dose BAY94-8862 IR tablet 1.25mg
  Interventions: Drug: BAY94-8862 (1.25mg)
- BAY94-8862 (2.5mg) (Experimental): single dose BAY94-8862 IR tablet 2.5mg
  Interventions: Drug: BAY94-8862 (2.5mg)
- BAY94-8862 (5mg) (Experimental): single dose BAY94-8862 IR tablet 5mg
  Interventions: Drug: BAY94-8862 (5mg)
- BAY94-8862 (7.5mg) (Experimental): single dose BAY94-8862 IR tablet 7.5mg
  Interventions: Drug: BAY94-8862 (7.5mg)
- BAY94-8862 (10mg) (Experimental): single dose BAY94-8862 IR tablet 10mg
  Interventions: Drug: BAY94-8862 (10mg)

INTERVENTIONS:
Drug: BAY94-8862 (1.25mg)
  Arms: BAY94-8862 (1.25mg)
Drug: BAY94-8862 (2.5mg)
  Arms: BAY94-8862 (2.5mg)
Drug: BAY94-8862 (5mg)
  Arms: BAY94-8862 (5mg)
Drug: BAY94-8862 (7.5mg)
  Arms: BAY94-8862 (7.5mg)
Drug: BAY94-8862 (10mg)
  Arms: BAY94-8862 (10mg)

SUMMARY:
This study should estimate the dose proportionality of BAY94-8862 IR tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 46 years (inclusive) at the first screening examination
* Ethnicity: White
* Body mass index (BMI): >= 18 and <= 29.9 kg / m²

Exclusion Criteria:

* Clinically relevant findings in the ECG (electrocardiogram) such as a second- or third-degree AV block, prolongation of the QRS complex over 120 msec
* Systolic blood pressure below 100 or above 140 mmHg
* Diastolic blood pressure below 50 or above 90 mmHg
* Heart rate below 50 or above 95 beats/ min
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus antibodies (anti-HIV 1+2)
* Participation in another clinical study during the preceding 3 months (Last Treatment from previous study to First Treatment of new study)

Ages: 18 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2012-11-28 (Actual); Study Completion 2013-03-21 (Actual)

PRIMARY OUTCOMES:
Dose proportionality of BAY94-8862 exposure in plasma when given as 1.25, 2.5, 5.0, 7.5 and 10 mg IR tablets | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 28 & 48 h

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of BAY94-8862 | Up to 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical-Research-Services Mönchengladbach GmbH, Mönchengladbach, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/